CLINICAL TRIAL: NCT06428539
Title: T Regulatory Cells in Lupus Nephritis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed AbdEllah Ahmed Hussein, Principal Investigator, Assiut University
Other Study IDs: T cells in lupus LN
Record Dates: First submitted 2024-05-21; First posted 2024-05-24 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients with active lupus nephritis: patients with active lupus nephritis as active urinary sediment, or rising renal chemistry
  Interventions: Diagnostic Test: T-reg cells
- patients with lupus nephritis in remission: Patients who were previously active, but now in remission
  Interventions: Diagnostic Test: T-reg cells
- normal individuals: normal healthy participants
  Interventions: Diagnostic Test: T-reg cells

INTERVENTIONS:
Diagnostic Test: T-reg cells — laboratory test
  Other Names: t regulatory cells

SUMMARY:
* To study the role FoxP3-positive T regulatory cells in the pathogenesis of Lupus Nephritis, and determine the factors associated with levels of T regs .
* To compare the functional capacity of T regs in LN and in normal individuals.

DETAILED DESCRIPTION:
Lupus Nephritis (LN) encompasses a group of glomerulonephrites, that occur in association with systemic lupus erythematosus (SLE). The mainstream theory that it is an immune disease resulting from loss of immune tolerance against body cells. The regulatory T cells (T regs ) are a subpopulation of immune cells that maintain tolerance to self-antigens and suppress autoimmune diseases. The main marker of Tregs is FoxP3 (forkhead box protein 3) positivity. Moreover, It has been suggested that functional capacity of Tregs is also compromised in autoimmune diseases. Studying the role of T regs in LN is a promising field that can help tailor current immune therapy and develop new treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

adults both genders clinical diagnosis of lupus nephritis

Exclusion Criteria:

patients diagnosed with other renal pathologies, e.g. diabetic kidney disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with lupus nephritis, both currently active or in remission, divided in Group 1: active lupus nephritis, Group 2: lupus nephritis in remission. Besides including normal Group 3: healthy volunteers
Sampling Method: Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
FoxP3 between groups | baseline
  mean difference of FoxP3 between groups.
Association of FoxP3 and activity index | baseline
  correlation between level of FoxP3 and activity index in the group with active LN.
Tregs in normal and lupus participants | baseline
  mean difference of suppression capacity of Tregs between normal participants and patients with active LN.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Doglio M, Alexander T, Del Papa N, Snowden JA, Greco R; Autoimmune Diseases Working Party (ADWP) of the European Society for Blood and Marrow Transplantation (EBMT). New insights in systemic lupus erythematosus: From regulatory T cells to CAR-T-cell strategies. J Allergy Clin Immunol. 2022 Dec;150(6):1289-1301. doi: 10.1016/j.jaci.2022.08.003. Epub 2022 Sep 20. PMID 36137815